CLINICAL TRIAL: NCT05129202
Title: Outcomes With Immune Checkpoint Inhibitor for Patients With Non-Small-Cell Lung Cancer and Stable Brain Metastases：A Retrospective Study
Brief Title: Outcomes With Immune Checkpoint Inhibitor for Patients With Non-Small-Cell Lung Cancer and Stable Brain Metastases
Acronym: OMESIA
Status: Completed | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Other Study IDs: OMESIA
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy, Active

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemotherapy alone or chemotherapy combined with anti-angiogenesis: patients with Chemotherapy
- immuntherapy: patients treated with immune checkpoint inhibitor monotherapy or combination therapy.
  Interventions: Drug: immune therapy

INTERVENTIONS:
Drug: immune therapy — The patient receives immunotherapy
  Groups: immuntherapy

SUMMARY:
Non-small cell lung cancer patients may have brain metastases at diagnosis. Patients with brain metastasis may contribute as poor prognosis factors. This trial aims to explore the efficacy and the safety of immune checkpoint inhibitors in non small cell lung cancer patients with initial brain metastasis.

ELIGIBILITY:
Inclusion Criteria:

* 1.Diagnosed with advanced non-small cell lung cancer 2.Patients with brain metastasis 3. Treated with ICIs

Exclusion Criteria:

* 1.Patients with a clear driver mutation that can be targeted for first-line treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain metastasis received immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
ORR | November 2017- October 2021
  disease remission rate
PFS | November 2017- October 2021
  progression free survival

SECONDARY OUTCOMES:
OS | November 2017- October 2021
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang C Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Huang Z, Wu F, Xu Q, Song L, Zhang X, Wang Z, Deng L, Zhang Y, Zeng L, Yang N. Intracranial activity of first-line immune checkpoint inhibitors combined with chemotherapy in advanced non-small cell lung cancer. Chin Med J (Engl). 2023 Jun 20;136(12):1422-1429. doi: 10.1097/CM9.0000000000002720. Epub 2023 May 17. PMID 37195128